CLINICAL TRIAL: NCT02289989
Title: Investigator-Initiated, Randomized, Investigator-Blind, Half-Side Comparison of Topical Oregano Extract Ointment vs .Hydrocortisone 1% for the Treatment of Atopic Dermatitis in Pediatric Patients
Brief Title: Oregano Ointment vs. Standard Treatment for Pediatric Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of response to recruitment
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2012002449
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Oregano; Atopic Dermatitis Quick (ADQ) score; Eczema Area and Severity Index score; Reflectance confocal microscopy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard: Hydrocortisone 1% ointment (Active Comparator): Intervention: hydrocortisone 1% ointment will be applied to one patient's forearm
  Interventions: Drug: Hydrocortisone
- Experimental: oregano extract cream (Experimental): Intervention: Oregano extract cream for mild to moderate atopic dermatitis will be applied to the other patient's forearm
  Interventions: Drug: Oregano extract cream

INTERVENTIONS:
Drug: Oregano extract cream — An experimental cream will be applied to one of the arms of the patient which will be an oregano extract and will be compared to the standard treatment which will be hydrocortisone 1% ointment
  Other Names: experimental treatment
  Arms: Experimental: oregano extract cream
Drug: Hydrocortisone — An experimental cream will be applied to one of the arms of the patient which will be an oregano extract and will be compared to the standard treatment which will be hydrocortisone 1% ointment
  Other Names: active control
  Arms: Standard: Hydrocortisone 1% ointment

SUMMARY:
This study is designed to evaluate and compare the efficacy of 3% oregano extract ointment prepared in aqueous solution versus 1% hydrocortisone ointment, a standard treatment, in decreasing the inflammation associated with mild to moderate atopic dermatitis. We plan to recruit 40 patients on the ages comprised between 2 and 17 years old and the study duration for each of the patient is 1 month.

DETAILED DESCRIPTION:
A single-center, investigator initiated, randomized controlled, double-blind trial will be conducted to determine the effects of an oregano extract in aqueous solution versus 1% hydrocortisone in the treatment of acute-subacute pediatric atopic dermatitis (AD). We suspect that topical oregano will serve as an effective, non-steroidal AD therapy, simultaneously offering extra benefits to pediatric patients as oregano is a natural product with antimicrobial, anti-inflammatory, and antiseptic properties that lacks reports of adverse effects associated with steroids, which children have been noted to be more susceptible to.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects aged 2-17 years of age.
* Individuals must be diagnosed with acute-subacute AD regardless of the study.
* Written informed consent must be obtained from all patients or caregivers.
* Women of childbearing potential (WOCBP) must be willing to practice effective contraception for the duration of study treatment.
* Subjects must be willing and able to comply with study conditions, properly apply or have caregivers apply topical medications to the selected body sites, as well as return to the clinic for required visits.
* Subject caregivers must be willing and able to perform ADQ assessment test.

Exclusion Criteria:

* Individuals who are immune-compromised or suffering from infectious disease, malignant disease, are known to be HIV+ or present with a general reduced level of health.
* Individuals diagnosed with underlying dermatological conditions in addition to AD.
* Individuals with a chronic pre-existing disease such as diabetes mellitus or others that in the opinion of the investigator would preclude their participation in the study.
* Individuals who are pregnant, nursing mothers, or subjects planning a pregnancy during the course of the study.
* Subjects/caregivers who are unable to communicate or comply with study conditions due to language disability, poor mental development, or impaired cerebral function.
* Individuals who are simultaneously enrolled in another clinical drug or device research study.
* Individuals with a history of chronic steroid use.
* Individuals needing to concurrently use topical agents, medicinal products containing corticosteroids, or immunosuppressants.
* Individuals who have received systemically administered corticosteroids and/or antihistamines 2 weeks prior to the start of study.
* Individuals undergoing light therapy.
* Individuals who have been treated with another investigation device or drug within 30 days prior to study enrollment.
* Individuals with a known allergy to oregano.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Pappert, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Department of Dermatology. Rutgers-RWJMS, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done in the department of dermatology of Rutgers-RWJMS. It was stopped in July 2016.
Pre-assignment Details: No exclusions or significant events were observed in the study.
Period: Overall Study
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Clinical Efficacy Rated by the Patient or Caregiver on Days 0 and 25
Description: This was measured with two questions. The first one referred to the description of the lesion and it included six characteristics: clear, dry, scaly, redness, cracks/opening and oozing. The second questions asked to grade how itchy was the patient.
  All characteristics were measured on a scale from 0 to 5 (0 none, 5 extremely bothered/losing sleep).
Time Frame: From baseline to day 25
Measure: Number; unit: participants
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 1
participants
  Scaly, redness, cracks/opening day 0 |  | 1
  Very bothered (4) day 0 |  | 1
  Scaly, Redness day 25 |  | 1
  Quite bothered (3) day 25 |  | 1

2. Primary Outcome: Change of the Clinical Efficacy Rated by a Study Physician
Description: Physician was asked to grade four characteristics: erythema, infiltration/papulation, excoriation and lichenification. The grade was none (0), mild (1), moderate (2) and severe (3).
Time Frame: Baseline to day 28
Measure: Number; unit: participants
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 1
participants
  Erythema day 0 severe |  | 1
  Infiltration/Papulation day 0 none |  | 1
  Excoriation day 0 severe |  | 1
  Lichenification day 0 moderate |  | 1
  Erythema day 28 moderate |  | 1
  Infiltration/Papulation day 28 none |  | 1
  Excoriation day 28 mild |  | 1
  Lichenification day 28 mild |  | 1

3. Primary Outcome: Histological Improvement Measured by Confocal Microscopy
Description: Confocal microscopy was done to the patient on day 0, day 14 and day 28. Due to technical difficulties, this outcome measure was not collected.
Time Frame: Baseline to day 28
Population: Data not collected
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measure Presence of S. Aureus Colonization on Affected Skin
Description: Bacterial culture of the affected area was done on day 0 and day 14.
Time Frame: Baseline to day 14
Measure: Number; unit: participants
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 1
participants
  Bacterial culture day 0 negative |  | 1
  Bacterial culture day 14 negative |  | 1

5. Secondary Outcome: Rate Cosmetic Acceptability of Topical Agents
Description: The patient or caregiver rated how the product felt on their skin after applying the product, measuring the cosmetic acceptability on day 7 and 14. The scale was excellent, good, moderate and poor.
Time Frame: On day 7 and 14
Measure: Number; unit: participants
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 1
participants
  Cosmetic acceptability day 7 excellent |  | 1
  Cosmetic acceptability day 14 excellent |  | 1

6. Secondary Outcome: Rate Skin Tolerance of Topical Agents
Description: The patient or caregiver rated how well the patient tolerated the product after applying it on day 7 and 14. The scale was excellent, good, moderate and poor.
Time Frame: On day 7 and 14
Measure: Number; unit: participants
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
Number analyzed (Participants) | 0 | 1
participants
  Skin tolerance day 7 excellent |  | 1
  Skin tolerance day 14 excellent |  | 1

ADVERSE EVENTS:
Arm/Group | Standard: Hydrocortisone 1% Ointment | Experimental: Oregano Extract Cream
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Termination of the trial due to difficulty recruiting patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No